CLINICAL TRIAL: NCT03357471
Title: A Multicenter, Open-Label Study to Evaluate the Safe and Effective Use of an Electro-Mechanical Injection Device (E-Device) for the Subcutaneous Self-Injection of Certolizumab Pegol Solution by Subjects With Moderate to Severe Active Rheumatoid Arthritis, Active Ankylosing Spondylitis, Active Psoriatic Arthritis, or Moderately to Severely Active Crohn's Disease
Brief Title: Study to Test the Safe and Effective Use of an e-Device for the Self-injection of Certolizumab Pegol Solution by Subjects With Moderate to Severe Active Rheumatoid Arthritis, Active Ankylosing Spondylitis, Active Psoriatic Arthritis, or Moderately to Severely Active Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RA0098
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2017-11-23; First posted 2017-11-30 (Actual); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Moderate and Severe Active Rheumatoid Arthritis; Active Psoriatic Arthritis; Active Ankylosing Spondylitis; Moderately to Severely Active Crohn's Disease
Keywords: Certolizumab Pegol; E-Device
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Certolizumab Pegol Q2W injection by e-Device (Experimental): Subjects will self-inject Certolizumab Pegol 200 mg (1 x 200 mg injection) using the e-Device every 2 weeks.
  Interventions: Drug: e-Device
- Certolizumab Pegol Q4W injection by e-Device (Experimental): Subjects will self-inject Certolizumab Pegol 400 mg (2 x 200 mg injection) using the e-Device every 4 weeks.
  Interventions: Drug: e-Device

INTERVENTIONS:
Drug: e-Device — * Active Substance: Certolizumab Pegol
  * Pharmaceutical form: Solution for injection
  * Route of administration: subcutaneous injection by e-Device
  Other Names: Cimzia

SUMMARY:
The purpose of the study is to evaluate the ability of subjects who are already prescribed Certolizumab Pergol therapy and have been self injecting with prefilled syringes for at least the previous three months, to safely and effectively self-inject Certolizumab Pegol (CZP) using the e-Device and to evaluate the post-use structural integrity of used devices and cassettes via visual examination.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and must be at least 18 years old at Visit 1
* Subject must have been diagnosed at least 6 months prior to Visit 1 with documented moderate to severe active Rheumatoid Arthritis (RA), active Psoriatic Arthritis (PsA), active Ankylosing Spondylitis (AS) (in US), or moderately to severely active Crohn's Disease (CD) (in US)
* A minimum of 10 subjects will have impaired hand function. Impaired hand function will be measured using the Cochin scale (Duruöz et al, 1996; Poiraudeau et al, 2000) and impaired hand function will be defined as patients who have a Cochin score >= 13.5 at Baseline
* Subjects must have been prescribed Certolizumab Pegol (CZP) and must have been self-injecting CZP using the pre-filled syringe for at least 3 months prior to Visit 1. Subjects with RA, PsA, or AS must have been on a stable Q2W (every 2 weeks) or Q4W (every 4 weeks) CZP dosing regimen for at least 3 months prior to Screening. Subjects with CD must have been on a stable Q4W CZP dosing regimen for at least 3 months prior to Visit 1.
* Subjects must have been screened according to the applicable national tuberculosis (TB) screening guidelines (to be documented) or provide a documented TB screening activity (TB questionnaire, Interferon-Gamma-Release Assay (IGRA) test, or chest x-ray) within the past 12 months prior to Visit 1.
* Female subjects of childbearing potential should have a negative pregnancy test at Visit 1 and should be using a medically accepted method of contraception during the entire duration of the study. Female subjects who are postmenopausal for at least 2 years or have undergone a complete hysterectomy, bilateral tubal ligation, and/or bilateral oophorectomy, or have a congenital sterility are considered not of childbearing potential

Exclusion Criteria:

* Subject has participated in another study of an investigational medicinal product (IMP) or an investigational device within the previous 3 months or is currently participating in another study of an IMP or an investigational device
* Subject has a history of chronic alcohol or drug abuse within the previous 6 months
* Subject has a history of significant cardiovascular, respiratory, gastrointestinal, hepatic, endocrine, renal, dermatological, neurological, psychiatric, hematological, or bleeding disorders
* Subjects with known Tuberculosis (TB) infection and at high risk of acquiring TB infection. Subjects with latent TB (LTB) who have not completed the prophylactic treatment regimen for LTB 3 months prior to enrollment
* Subject has an active chronic/latent infection including but not limited to TB (untreated latent or active), hepatitis virus (HV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
* Subject has a current malignancy or a history of malignancy. Subjects with less than 3 completely excised basal cell carcinomas or with cervical carcinoma in situ successfully treated surgically more than 5 years prior to Screening may be included
* Subject has had major surgery (including joint surgery) within 8 weeks prior to Visit 1, or has a scheduled surgery during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (22):
- United States (22):
  - Ra0098 116, Mesa, Arizona
  - Ra0098 107, Mesa, Arizona
  - Ra0098 135, Phoenix, Arizona
  - Ra0098 119, Tucson, Arizona
  - Ra0098 101, Covina, California
  - Ra0098 131, Clermont, Florida
  - Ra0098 132, Coral Springs, Florida
  - Ra0098 127, Gainesville, Georgia
  - Ra0098 122, Clive, Iowa
  - Ra0098 105, St Louis, Missouri
  - Ra0098 104, St Louis, Missouri
  - Ra0098 103, Dover, New Jersey
  - Ra0098 117, Great Neck, New York
  - Ra0098 113, Myrtle Beach, South Carolina
  - Ra0098 126, Hixson, Tennessee
  - Ra0098 111, Austin, Texas
  - Ra0098 123, Austin, Texas
  - Ra0098 102, Austin, Texas
  - Ra0098 128, Corpus Christi, Texas
  - Ra0098 106, Nassau Bay, Texas
  - Ra0098 114, San Antonio, Texas
  - Ra0098 133, Richland, Washington

REFERENCES:
- [Derived] Pompilus F, Ciesluk A, Strzok S, Ciaravino V, Harris K, Szegvari B, Mountian I, Cleanthous S, Meunier J. Development and psychometric evaluation of the assessment of self-injection questionnaire: an adaptation of the self-injection assessment questionnaire. Health Qual Life Outcomes. 2020 Nov 4;18(1):355. doi: 10.1186/s12955-020-01606-7. PMID 33148261
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in November 2017 and concluded in July 2018.
Pre-assignment Details: Participant Flow refers to the Safety Set (SS), which consisted of all subjects of the study who had received at least 1 dose of CZP during the study (e-Device).
Groups:
- Certolizumab Pegol Q2W Injection by e-Device: Subjects self-injected Certolizumab Pegol 200 mg (1 x 200 mg injection) using the e-Device every 2 weeks.
- Certolizumab Pegol Q4W Injection by e-Device: Subjects self-injected Certolizumab Pegol 400 mg (2 x 200 mg injection) using the e-Device every 4 weeks.
Period: Overall Study
Arm/Group | Certolizumab Pegol Q2W Injection by e-Device | Certolizumab Pegol Q4W Injection by e-Device
Started | 35 | 32
Completed | 33 | 32
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refers to the Safety Set which consisted of all subjects who received at least 1 dose of CZP during the study (e-Device).
Arm/Group | Certolizumab Pegol Q2W Injection by e-Device | Certolizumab Pegol Q4W Injection by e-Device | Total Title
Number analyzed (Participants) | 35 | 32 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 24 | 53
  >=65 years | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (13.1) | 52.6 (13.6) | 52.4 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 14 | 7 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Black | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 33 | 30 | 63
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Able to Self-administer Safe and Effective Injections Using the e-Device at Visit 2
Description: Safe and effective self-injection was evaluated by the healthcare provider and is defined as:
  * Dose Delivery: Subject self-injected the complete dose of Certolizumab Pegol (CZP) as confirmed by a visual inspection of the CZP-cassette(s) which shows the pre-filled syringe container to be empty AND
  * No Adverse Events related to use of the e-Device (Adverse Device Effects) that would preclude continued use of the e-Device for self-injection.
  For subjects on the Q4W (every 4 weeks) dosing regimen who would self-inject twice (2×200 mg CZP) at each visit, each injection was evaluated for safety and effectiveness using the above criteria. The primary endpoint of safe and effective self-injection for subjects on the Q4W dosing regimen was met only if both self-injections were determined to be safe and effective.
Time Frame: Visit 2 (Week 2 for Q2W; Week 4 for Q4W)
Population: The Safety Set (SS) consisted of all subjects of the study who had received at least 1 dose of CZP during the study (e-Device). Percentages were based on the number of SS subjects that participated in Visit 2 and received at least 1 dose of CZP.
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Groups:
- Certolizumab Pegol Q2W Injection by e-Device (SS): Subjects self-injected Certolizumab Pegol 200 mg (1 x 200 mg injection) using the e-Device every 2 weeks. Subjects formed the Safety Set (SS).
- Certolizumab Pegol Q4W Injection by e-Device (SS): Subjects self-injected Certolizumab Pegol 400 mg (2 x 200 mg injection) using the e-Device every 4 weeks. Subjects formed the Safety Set (SS).
Arm/Group | Certolizumab Pegol Q2W Injection by e-Device (SS) | Certolizumab Pegol Q4W Injection by e-Device (SS)
Number analyzed (Participants) | 33 | 32
percentage of subjects | 100.00 [91.3 to 100.0] | 96.88 [86.0 to 99.8]

2. Secondary Outcome: Percentage of Subjects Able to Self-administer Safe and Effective Injections Using the e-Device at Visit 1
Description: as for outcome 1
Time Frame: Visit 1 (Week 0)
Population: The Safety Set (SS) consisted of all subjects of the study who had received at least 1 dose of CZP during the study (e-Device). Percentages were based on the number of SS subjects that participated in Visit 1 and received at least 1 dose of CZP.
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol Q2W Injection by e-Device (SS) | Certolizumab Pegol Q4W Injection by e-Device (SS)
Number analyzed (Participants) | 35 | 32
percentage of subjects | 100.00 [91.8 to 100.0] | 100.00 [91.1 to 100.0]

3. Secondary Outcome: Percentage of Used Certolizumab Pegol (CZP)-Cassettes Identified as Having Structural Integrity Issues Based on Visual Examination
Description: CZP-cassettes identified as having structural integrity issues meant CZP-cassettes with clear evidence of damage/compromised structural integrity, not superficial cosmetic imperfections.
Time Frame: During the study (from Week 0 up to Week 4)
Population: The Safety Set (SS) consisted of all subjects of the study who had received at least 1 dose of CZP during the study (e-Device). Percentages were based on the number of cassettes evaluated.
Measure: Number (90% Confidence Interval); unit: percentage of cassettes
Units Other Than Participants: CZP - cassettes
Arm/Group | Certolizumab Pegol Q2W Injection by e-Device (SS) | Certolizumab Pegol Q4W Injection by e-Device (SS)
Number analyzed (Participants) | 35 | 32
Number analyzed (CZP - cassettes) | 68 | 128
percentage of cassettes | 0 [0.0 to 4.3] | 0 [0.0 to 2.3]

4. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure
Description: Blood pressure was measured in millimetre of mercury (mmHg).
Time Frame: From Week 0 to Visit 2 (Week 2 for Q2W; Week 4 for Q4W)
Population: The Safety Set (SS) consisted of all subjects of the study who had received at least 1 dose of CZP during the study (e-Device). The mean was based on the number of SS subjects that participated in Visit 2 and received at least 1 dose of CZP.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Certolizumab Pegol Q2W Injection by e-Device (SS) | Certolizumab Pegol Q4W Injection by e-Device (SS)
Number analyzed (Participants) | 33 | 32
mmHg | -0.12 (9.04) | -2.31 (10.98)

5. Secondary Outcome: Mean Change From Baseline in Diastolic Blood Pressure
Description: Blood pressure was measured in millimetre of mercury (mmHg).
Time Frame: From Week 0 to Visit 2 (Week 2 for Q2W; Week 4 for Q4W)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Certolizumab Pegol Q2W Injection by e-Device (SS) | Certolizumab Pegol Q4W Injection by e-Device (SS)
Number analyzed (Participants) | 33 | 32
mmHg | -1.21 (7.03) | -2.25 (10.24)

6. Secondary Outcome: Mean Change From Baseline in Pulse Rate
Description: Pulse Rate was measured in beats per minute (beats/min).
Time Frame: From Week 0 to Visit 2 (Week 2 for Q2W; Week 4 for Q4W)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Certolizumab Pegol Q2W Injection by e-Device (SS) | Certolizumab Pegol Q4W Injection by e-Device (SS)
Number analyzed (Participants) | 33 | 32
beats/min | -0.42 (6.45) | -0.97 (9.32)

7. Secondary Outcome: Mean Change From Baseline in Respiratory Rate
Description: Respiratory Rate was measured in breaths per minute (breaths/min).
Time Frame: From Week 0 to Visit 2 (Week 2 for Q2W; Week 4 for Q4W)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Certolizumab Pegol Q2W Injection by e-Device (SS) | Certolizumab Pegol Q4W Injection by e-Device (SS)
Number analyzed (Participants) | 33 | 32
breaths/min | -0.48 (1.73) | -0.19 (2.18)

8. Secondary Outcome: Mean Change From Baseline in Body Temperature
Description: Body Temperature was measured in Grad Celsius (°C).
Time Frame: From Week 0 to Visit 2 (Week 2 for Q2W; Week 4 for Q4W)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Temperature (C)
Arm/Group | Certolizumab Pegol Q2W Injection by e-Device (SS) | Certolizumab Pegol Q4W Injection by e-Device (SS)
Number analyzed (Participants) | 33 | 32
Temperature (C) | 0.05 (0.41) | -0.06 (0.34)

9. Secondary Outcome: Incidence of Adverse Events (AEs) During the Study
Description: An Adverse Event (AE) was any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of investigational medicinal product (IMP), whether or not related to the medicinal (investigational) product.
Time Frame: During the study (from Week 0 up to Week 5 +/-3 Days)
Population: The Safety Set (SS) consisted of all subjects of the study who had received at least 1 dose of CZP during the study (e-Device).
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol Q2W Injection by e-Device (SS) | Certolizumab Pegol Q4W Injection by e-Device (SS)
Number analyzed (Participants) | 35 | 32
percentage of participants | 14.3 | 12.5

10. Secondary Outcome: Incidence of Adverse Device Events (ADEs) During the Study
Description: An Adverse Device Event (ADE) was an AE related to the use of an investigational device. An ADE must have met 1 or more of the following criteria:
  * Adverse event that resulted from insufficiencies or inadequacies in the Instructions for Use (IFU), the deployment, the implantation, the installation, the operation, or any malfunction of the investigational medical device
  * Adverse event that was a result of an error or intentional misuse.
Time Frame: During the study (from Week 0 up to Week 5 +/-3 Days)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol Q2W Injection by e-Device (SS) | Certolizumab Pegol Q4W Injection by e-Device (SS)
Number analyzed (Participants) | 35 | 32
percentage of participants | 0 | 3.1

ADVERSE EVENTS:
Time Frame: From the start of Treatment Period at Week 0 and up to Safety Follow-Up (1 week after the subject's final site visit using the e-Device), an average of 5 Weeks +/-3 Days.
Arm/Group | Certolizumab Pegol Q2W Injection by e-Device (SS) | Certolizumab Pegol Q4W Injection by e-Device (SS)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/32
Other Adverse Events (participants affected / at risk) | 0/35 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT03357471/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT03357471/SAP_001.pdf